CLINICAL TRIAL: NCT05024513
Title: Prospective Multicentre Trial of Biliary Drainage Plus Hepatic Arterial Infusion Chemotherapy Versus Biliary Drainage Plus Best Supportive Care in Locally Advanced Perihilar Cholangiocarcinomas.
Brief Title: Biliary Drainage Plus HAIC in Locally Advanced pCCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAIC
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: Perihilar Cholangiocarcinoma; Hepatic arterial infusion chemotherapy; Biliary Drainage; Best Supportive Care
MeSH Terms: conditions — Klatskin Tumor | interventions — Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BD-HAIC (Biliary drainage & HAIC) (Experimental): The patients enrolled in this arm would receive external percutaneous biliary drainage plus 3Cir-OFF hepatic arterial infusion chemotherapy （HAIC）with oxaliplatin and 5-fluorouracil.
  Interventions: Drug: oxaliplatin and 5-fluorouracil; Procedure: External biliary drainage
- BD-BSC (Biliary Drainage & Best supportive care) (Active Comparator): The patients enrolled in this arm would receive biliary drainage, biliary stents,or biliary stents with Iodine-125 seed strands, plus best supportive care.
  Interventions: Procedure: Biliary Drainage; Other: Best Supportive Care

INTERVENTIONS:
Drug: oxaliplatin and 5-fluorouracil — Intra-arterial chemotherapy consisted of Oxaliplatin (40mg/m2 for 2 hours), 5-fluorouracil (800 mg/ m2 for22 hours) on days 1-3 every 4 weeks.
  Arms: BD-HAIC (Biliary drainage & HAIC)
Procedure: Biliary Drainage — External biliary drainage, or biliary stent placement; Biliary stent placement plus Iodine-125 seed strands is allowed
  Arms: BD-BSC (Biliary Drainage & Best supportive care)
Other: Best Supportive Care — Nutrition support, symptomatic treatment, and other supportive treatments
  Arms: BD-BSC (Biliary Drainage & Best supportive care)
Procedure: External biliary drainage — External biliary drainage
  Arms: BD-HAIC (Biliary drainage & HAIC)

SUMMARY:
Biliary drainage and stent placement remains to be the main palliative treatment choice for advanced perihiliar cholangiocarcinoma (pCCA), and the life expectancy is only 4-6 months. Previous single center prospective phase 2 trial showed that hepatic arterial infusion chemotherapy (HAIC) with oxaliplatin and 5-fluorouracil was an encouraging treatment choice for advanced pCCA due to its high tumor control, survival benefit, and low toxicity. Thus, the multicenter prospective controlled trial was designed to explore and confirm the survival benefit of biliary drainage plus hepatic arterial infusion chemotherapy with oxaliplatin and 5-fluorouracil compared with biliary drainage plus best support care treatment in locally advanced pCCA patients.

DETAILED DESCRIPTION:
When a patient is not eligible for surgery, chemotherapy with gemcitabine and cisplatin can be considered for advanced biliary tract cancer. However, in the Advanced Biliary Tract Cancer, or ABC-02 trial in patients with pCCA, the efficacy of this regimen was not significantly higher than that of gemcitabine alone. Therefore, an optimal chemotherapeutic regimen has not been established for this subtype of cholangiocarcinoma. Currently, biliary drainage and stent placement remains to be the main palliative treatment choice, and the life expectancy is only 4-6 months. Previous single center prospective phase 2 trial showed that HAI with oxaliplatin and 5-fluorouracil was an encouraging treatment choice for advanced PCC due to its high tumor control, survival benefit, and low toxicity. So the multicenter prospective controlled trial was designed to explore and confirm the survival benefit of biliary drainage plus hepatic arterial infusion of oxaliplatin and 5-fluorouracil compared with biliary drainage plus best support care treatment in locally advanced pCCA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced perihilar cholangiocarcinoma proved by histology or cytology.
2. Locally advanced unresectable perihilar cholangiocarcinoma, decided by hepatobiliary doctor and radiologist.
3. Age from 18 years old to 80 years old.
4. The performance of Eastern Cooperative Oncology Group (ECOG) <2
5. Child-Pugh A or Child-Pugh B (≤ grade 7).
6. Expectant survival time ≥ 3 months.
7. Baseline blood count test and blood biochemical must meet following criteria:

   1. Hemoglobin ≥ 90 g/L;
   2. Absolute neutrophil count ≥ 1.5×10^9/L;
   3. Blood platelet count ≥ 100×10^9/L;
   4. Serum creatinine ≤ 1.5 times of ULN;
   5. Albumin ≥ 30 g/L
8. Patients sign informed consent.

Exclusion Criteria:

1. Allergic to contrast agent.
2. Pregnant or lactational.
3. Allergic to 5-fluorouracil, or have metabolic disorder of 5-fluorouracil.
4. Previous systematic chemotherapy or radiotherapy.
5. Patients with complications such as bile leakage and bleeding after PTCD
6. N2 lymphatic metastasis, extrahepatic metastasis, or coinstantaneous a lot of malignant hydrothorax or ascites.
7. History of organ transplantation.
8. Coinstantaneous infection and need anti-infection therapy.
9. Coinstantaneous peripheral nervous system disorder or with history of obvious mental disorder and central nervous system disorder.
10. Diagnosed other kinds of malignant within 5 years, except for non-melanoma skin cancer and carcinoma in situ of cervix.
11. Without legal capacity.
12. Uncorrectable coagulation disorder.
13. Obvious abnormal in ECG or obvious clinical symptoms of heartdisease, like congestive heart failure (CHF), coronary heart disease with obvious clinical symptoms, unmanageable arrhythmia and hypertension.
14. Severe liver disease (like cirrhosis), renal disease, respiratory disease,unmanageable diabetes or other kinds of systematic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Overall survival is measured from the date of first biliary drainage to death

SECONDARY OUTCOMES:
Duration of jaundice remission | 1 year
  The time between remission of total bilirubin to less than 2 times of the upper limit of the normal value and time of rising again of bilirubin above more than 2 times of upper limit of the normal level.

OTHER OUTCOMES:
Adverse effects | 6 months
  Toxicities were graded according to the Common Terminology Criteria for Adverse Events, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, Principal Investigator — Department of Interventional Oncology, Peking University Cancer Hospital
Locations (1):
- Department of Interventional Oncology, Key Laboratory of Carcinogenesis and Translational Research (Ministry of Education),Peking University Cancer Hospital and Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No
signed informed consent with patients

REFERENCES:
- [Background] Ilyas SI, Khan SA, Hallemeier CL, Kelley RK, Gores GJ. Cholangiocarcinoma - evolving concepts and therapeutic strategies. Nat Rev Clin Oncol. 2018 Feb;15(2):95-111. doi: 10.1038/nrclinonc.2017.157. Epub 2017 Oct 10. PMID 28994423
- [Background] Banales JM, Cardinale V, Carpino G, Marzioni M, Andersen JB, Invernizzi P, Lind GE, Folseraas T, Forbes SJ, Fouassier L, Geier A, Calvisi DF, Mertens JC, Trauner M, Benedetti A, Maroni L, Vaquero J, Macias RI, Raggi C, Perugorria MJ, Gaudio E, Boberg KM, Marin JJ, Alvaro D. Expert consensus document: Cholangiocarcinoma: current knowledge and future perspectives consensus statement from the European Network for the Study of Cholangiocarcinoma (ENS-CCA). Nat Rev Gastroenterol Hepatol. 2016 May;13(5):261-80. doi: 10.1038/nrgastro.2016.51. Epub 2016 Apr 20. PMID 27095655
- [Background] Forner A, Vidili G, Rengo M, Bujanda L, Ponz-Sarvise M, Lamarca A. Clinical presentation, diagnosis and staging of cholangiocarcinoma. Liver Int. 2019 May;39 Suppl 1:98-107. doi: 10.1111/liv.14086. Epub 2019 Mar 25. PMID 30831002
- [Background] Nath MC, Torbenson MS, Erickson LA. Perihilar Cholangiocarcinoma. Mayo Clin Proc. 2018 Mar;93(3):397-398. doi: 10.1016/j.mayocp.2018.01.017. No abstract available. PMID 29502573
- [Background] Park J, Kim MH, Kim KP, Park DH, Moon SH, Song TJ, Eum J, Lee SS, Seo DW, Lee SK. Natural History and Prognostic Factors of Advanced Cholangiocarcinoma without Surgery, Chemotherapy, or Radiotherapy: A Large-Scale Observational Study. Gut Liver. 2009 Dec;3(4):298-305. doi: 10.5009/gnl.2009.3.4.298. Epub 2009 Dec 31. PMID 20431764
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Boehm LM, Jayakrishnan TT, Miura JT, Zacharias AJ, Johnston FM, Turaga KK, Gamblin TC. Comparative effectiveness of hepatic artery based therapies for unresectable intrahepatic cholangiocarcinoma. J Surg Oncol. 2015 Feb;111(2):213-20. doi: 10.1002/jso.23781. Epub 2014 Sep 1. PMID 25176325
- [Background] Hu J, Zhu X, Wang X, Cao G, Wang X, Yang R. Evaluation of percutaneous unilateral trans-femoral implantation of side-hole port-catheter system with coil only fixed-catheter-tip for hepatic arterial infusion chemotherapy. Cancer Imaging. 2019 Mar 18;19(1):15. doi: 10.1186/s40644-019-0202-z. PMID 30885278
- [Background] Wang X, Hu J, Cao G, Zhu X, Cui Y, Ji X, Li X, Yang R, Chen H, Xu H, Liu P, Li J, Li J, Hao C, Xing B, Shen L. Phase II Study of Hepatic Arterial Infusion Chemotherapy with Oxaliplatin and 5-Fluorouracil for Advanced Perihilar Cholangiocarcinoma. Radiology. 2017 May;283(2):580-589. doi: 10.1148/radiol.2016160572. Epub 2016 Nov 7. PMID 27820684